CLINICAL TRIAL: NCT00062140
Title: A Phase I Trial Of Total Body Irradiation, Cyclophosphamide Dose-Adjustment Based On Its Metabolism, And Hematopoietic Stem Cell Transplantation For Patients With Hematological Malignancy
Brief Title: Total-Body Irradiation, Cyclophosphamide, and Stem Cell Transplantation in Treating Patients With Hematologic Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: 1797.00; FHCRC-1797.00; CDR0000304522 (Registry Identifier: PDQ)
Record Dates: First submitted 2003-06-05; First posted 2003-06-06 (Estimated); Last update posted 2010-09-21 (Estimated); Status verified 2010-09

CONDITIONS: Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic/Myeloproliferative Diseases
Keywords: recurrent adult diffuse large cell lymphoma; recurrent adult diffuse mixed cell lymphoma; recurrent adult diffuse small cleaved cell lymphoma; recurrent adult Burkitt lymphoma; recurrent adult Hodgkin lymphoma; recurrent adult immunoblastic large cell lymphoma; recurrent adult lymphoblastic lymphoma; recurrent cutaneous T-cell non-Hodgkin lymphoma; recurrent grade 1 follicular lymphoma; recurrent grade 2 follicular lymphoma; recurrent grade 3 follicular lymphoma; recurrent mantle cell lymphoma; noncontiguous stage II adult diffuse large cell lymphoma; noncontiguous stage II adult diffuse mixed cell lymphoma; noncontiguous stage II adult Burkitt lymphoma; noncontiguous stage II adult immunoblastic large cell lymphoma; noncontiguous stage II adult lymphoblastic lymphoma; noncontiguous stage II grade 3 follicular lymphoma; noncontiguous stage II mantle cell lymphoma; stage III adult lymphoblastic lymphoma; stage IV adult lymphoblastic lymphoma; stage III adult Burkitt lymphoma; stage IV adult Burkitt lymphoma; recurrent adult acute myeloid leukemia; untreated adult acute myeloid leukemia; accelerated phase chronic myelogenous leukemia; blastic phase chronic myelogenous leukemia; chronic phase chronic myelogenous leukemia; meningeal chronic myelogenous leukemia; relapsing chronic myelogenous leukemia; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; noncontiguous stage II adult diffuse small cleaved cell lymphoma; noncontiguous stage II grade 1 follicular lymphoma; noncontiguous stage II grade 2 follicular lymphoma; recurrent mycosis fungoides/Sezary syndrome; secondary acute myeloid leukemia; stage III grade 1 follicular lymphoma; stage III grade 2 follicular lymphoma; stage III adult diffuse small cleaved cell lymphoma; stage III grade 3 follicular lymphoma; stage III adult diffuse large cell lymphoma; stage III adult diffuse mixed cell lymphoma; stage III adult immunoblastic large cell lymphoma; stage III mantle cell lymphoma; stage IV grade 3 follicular lymphoma; stage IV adult diffuse large cell lymphoma; stage IV adult diffuse mixed cell lymphoma; stage IV adult immunoblastic large cell lymphoma; stage IV mantle cell lymphoma; stage IV adult diffuse small cleaved cell lymphoma; stage IV grade 1 follicular lymphoma; stage IV grade 2 follicular lymphoma; recurrent adult acute lymphoblastic leukemia; untreated adult acute lymphoblastic leukemia; atypical chronic myeloid leukemia; myelodysplastic/myeloproliferative disease, unclassifiable; noncontiguous stage II small lymphocytic lymphoma; noncontiguous stage II marginal zone lymphoma; recurrent marginal zone lymphoma; recurrent small lymphocytic lymphoma; stage III small lymphocytic lymphoma; stage III marginal zone lymphoma; stage IV small lymphocytic lymphoma; stage IV marginal zone lymphoma; extranodal marginal zone B-cell lymphoma of mucosa-associated lymphoid tissue; nodal marginal zone B-cell lymphoma; splenic marginal zone lymphoma; adult acute myeloid leukemia with t(8;21)(q22;q22); adult acute myeloid leukemia with t(16;16)(p13;q22); adult acute myeloid leukemia with inv(16)(p13;q22); adult acute myeloid leukemia with 11q23 (MLL) abnormalities; adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Lymphoma; Myelodysplastic Syndromes; Myelodysplastic-Myeloproliferative Diseases; Lymphoma, Large B-Cell, Diffuse; Lymphoma, Non-Hodgkin; Burkitt Lymphoma; Hodgkin Disease; Lymphoma, Large-Cell, Immunoblastic; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Lymphoma, T-Cell, Cutaneous; Lymphoma, Follicular; Lymphoma, Mantle-Cell; Leukemia, Myeloid, Acute; Leukemia, Myeloid, Accelerated Phase; Blast Crisis; Leukemia, Myeloid, Chronic-Phase; Mycosis Fungoides; Sezary Syndrome; Leukemia, Myeloid, Chronic, Atypical, BCR-ABL Negative; Myeloproliferative Disorders; Lymphoma, B-Cell, Marginal Zone; Leukemia, Lymphocytic, Chronic, B-Cell; Congenital Abnormalities | interventions — Cyclophosphamide; Peripheral Blood Stem Cell Transplantation; Radiotherapy

INTERVENTIONS:
Drug: cyclophosphamide
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation
Radiation: radiation therapy

SUMMARY:
RATIONALE: Adjusting the dose of drugs used in chemotherapy such as cyclophosphamide may decrease side effects while stopping cancer cells from dividing so they stop growing or die. Radiation therapy uses high-energy x-rays to damage cancer cells. Stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy and radiation therapy used to kill cancer cells.

PURPOSE: Phase I trial to study the effect on the body of dose-adjusted cyclophosphamide combined with total-body irradiation and donor stem cell transplantation in treating patients who have hematologic cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine a safe and reproducible method of adjusting the dose of cyclophosphamide based on its metabolism when given in combination with total body irradiation and hematopoietic stem cell transplantation in patients with hematologic malignancy.

OUTLINE:

* Preparative regimen: Patients undergo total body irradiation twice daily on days -6 to -4. Patients then receive dose-adjusted (based on metabolism) cyclophosphamide IV over 1 hour on days -3 and -2.
* Hematopoietic stem cell (HSC) infusion: Patients undergo allogeneic HSC transplantation on day 0.

Patients receive graft-versus-host disease prophylaxis, CNS prophylaxis, and testicular irradiation as per institutional standard practices.

Patients are followed daily until day 80 after transplantation and then regularly thereafter for survival.

PROJECTED ACCRUAL: A total of 20 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of hematological malignancy, including any of the following:

  * Chronic myeloid leukemia
  * Acute myeloid leukemia
  * Acute lymphocytic leukemia
  * Myelodysplastic syndromes
  * Lymphoma
* Unlikely to respond to conventional treatment and would benefit from hematopoietic stem cell transplantation
* No bulky tumor mass requiring additional involved field radiotherapy
* No large body burden of tumor cells requiring cytoreductive chemotherapy before total body irraditation and cyclophosphamide
* Undergoing conditioning for transplantation at the University of Washington Medical Center
* Availability of 1 of the following types of allogeneic donors:

  * HLA-identical family members
  * Unrelated donors

    * Allele match (match grade 1)
    * One allele mismatch for A, B, C, DRB1 or DQB1 (match grades 2.1 or 2.2)

PATIENT CHARACTERISTICS:

Age

* 18 to 65

Performance status

* Not specified

Life expectancy

* Not severely limited by diseases other than malignancy
* Not moribund

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 1.2 mg/dL
* No cirrhosis
* No hepatic fibrosis with bridging

Renal

* Creatinine no greater than 1.2 mg/dL

Cardiovascular

* No coronary artery disease
* No congestive heart failure requiring therapy

Pulmonary

* Oxygen saturation at least 93% (on room air)

Other

* Not pregnant or nursing
* Fertile patients must use effective contraception
* HIV negative
* No concurrent infection requiring systemic antibiotic or antifungal therapy

PRIOR CONCURRENT THERAPY:

Biologic therapy

* No prior hematopoietic stem cell transplantation

Chemotherapy

* See Disease Characteristics

Endocrine therapy

* Not specified

Radiotherapy

* See Disease Characteristics
* No prior radiotherapy to the liver or adjacent organs

Surgery

* Not specified

Other

* No concurrent aspirin or nonsteroidal anti-inflammatory medications such as ibuprofen (e.g., Motrin® or Advil®)
* No other concurrent phase I study enrollment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2003-04; Study Completion 2004-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: George B. McDonald, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States